CLINICAL TRIAL: NCT06778109
Title: Manage Your Negative Thoughts: Stress, Anxiety Management Through Hypnosis in Medical Trainees
Brief Title: Manage Your Workingnegative Thoughts Through Hypnosis
Acronym: Hypnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Annalisa Boscolo, Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IPNOSIS
Record Dates: First submitted 2024-12-29; First posted 2025-01-16 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Stress; Stress Disorders
Keywords: stress; disorder; hypnosis
MeSH Terms: conditions — Stress Disorders, Traumatic; Disease | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypnosis and negative memory (Experimental): T0) basal evaluation of physiological data T1) evaluation of physiological data after recollecting a negative memory for 3 minutes T2) evaluation of physiological data after that a brief session of hypnosis (performed with positive memories) T3) evaluation of physiological data recolling, for the second time, the negative memory.
  Interventions: Other: hypnosis

INTERVENTIONS:
Other: hypnosis — T0) basal evaluation of physiological data T1) evaluation of physiological data after recollecting a negative memory for 3 minutes T2) evaluation of physiological data after that a brief session of hypnosis (performed with positive memories) T3) evaluation of physiological data recolling, for the second time, the negative memory.

SUMMARY:
Medical doctor generally are exposed to several risks and pressures, it is not a case that several meta-analyses have shown high stress and anxiety level in these workers. Stress management represents a very important topic. Being a doctor means dealing with continous effort and arousal management to provide the best treatment through executive functions capacity. This is particularly true for younger medical trainees; that have also to learn how to deal with failure and the curve of learning. Hypnosis has been shown to be very effective at modulating executive functions and sympathovagal balance, with large effect in post traumatic stress disease (PTSD), anxiety and executive function modulation. Therefore, this study aim to investigate if hypnosis could be beneficial among medical trainees for managing negative thoughts related to work.

DETAILED DESCRIPTION:
Stress and anxiety are very important issues in medical training. Several methods have been applied, from psychotherapy to biofeedback, but the physiological component usually have been dismissed. Training medical trainees to manage their physiological activity through hypnosis can probably transfer practical results, i.e. increased wellbeing, modulation of the working energy and the transfer from planning to properly execution. To obtain this results after a basal evaluation of physiological data (HR; Heart rate, HRV, Heart Rate Variability, EDA; Electrodermal activity, and SCr; Skin conductance responses) stress and of anxiety levels, , with PSS-10 scale, VAS stress, VAS anxiety and Tower of London test ( TOL-R), participants will recollect a negative memory for 3 minutes to monitor their response. After that a brief session of hypnosis will be performed with positive memories being recollected while all physiological data will be monitored. Then participants will be subjected again to the negative memory task end at the end of the session the same test of the basal evaluation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old,
* being medical doctor or at first year of residency in Anesthesiology
* obtained written informed consent

Exclusion Criteria:

* Neurological issues affecting stress responses
* Diabetes
* Cardiovascular conditions (i.e., hypertension, orthostatic hypotension etc)
* Being under psychiatric medications
* Psychological or psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the variations of the tonic and phasic component of the Electrodermal Activity (EDA,microSiemens) and Skin conductance response comparing pre and post-hypnosis (SCr/min) | T0) Within 3 minutes from electrodes application (at baseline), T1) within 3minute after a negative memory (w/o hypnosis), T2) within 3minutes after a positive memory, T3) within 3minutes after recalling the negative memory (after hypnosis application)
  Evaluation of the variations of the tonic and phasic component of the Electrodermal Activity (EDA,microSiemens) and Skin conductance response comparing pre and post-hypnosis (SCr/min)
Evaluation of the executive performance comparing pre- and post-hypnosis through Tower of London-Revised (TOL-R) (number of correct responses) | Within 3 minutes from the first negative memory (without hypnosis) and then, within 3 minutes from the negative memory (with hypnosis)
  Evaluation of the executive performance comparing pre- and post-hypnosis through Tower of London-Revised (TOL-R) (number of correct responses)

SECONDARY OUTCOMES:
Evaluation of the variations of psychological stress response to a negative memory related to work between pre and post hypnosis on a scale from 0 to 10 | Within 3 minutes from the first negative memory (without hypnosis) and then, within 3 minutes from the negative memory (with hypnosis)
  Evaluation of the variations of psychological stress response to a negative memory related to work between pre and post hypnosis on a scale from 0 to 10
Evaluation of the Heart rate variability (HRV) comparing pre and post-hypnosis (ms) | T0) Within 3 minutes from electrodes application (at baseline), T1) within 3minute after a negative memory (w/o hypnosis), T2) within 3minutes after a positive memory, T3) within 3minutes after recalling the negative memory (after hypnosis application)
  Evaluation of the Heart rate variability (HRV) comparing pre and post-hypnosis (ms)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto di Anestesia e Rianimazione, Padua, Italy
  - University of Padova, Padua, PD

IPD SHARING:
Plan to Share IPD: No